CLINICAL TRIAL: NCT04958655
Title: Estimating the Acute Impact of Competing Mental Imagery on Craving in Alcohol Use Disorder
Brief Title: Mental Imagery Intervention for Alcohol Craving
Acronym: ACLIMAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 295682
Record Dates: First submitted 2021-06-25; First posted 2021-07-12 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2021-06

CONDITIONS: Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetris, Positive Image (Other): Participants randomised to order of intervention: this arm has; Tetris (Active Comparator) then Positive Future Image (Intervention).
  Interventions: Behavioral: Tetris Task; Behavioral: Mental Imagery for Craving Reduction
- Positive Image, Tetris (Other): Participants randomised to order of intervention: this arm has; Positive Future Image (Intervention) then Tetris (Active Comparator).
  Interventions: Behavioral: Tetris Task; Behavioral: Mental Imagery for Craving Reduction

INTERVENTIONS:
Behavioral: Tetris Task — a visual task where participants are asked to play 'tetris' i.e. attend to and manipulate shapes and positions on screen
Behavioral: Mental Imagery for Craving Reduction — a behavioural mental imagery intervention where participants are asked to generate a specific future mental image to reduce cue-induced craving for alcohol

SUMMARY:
A within-subjects crossover, randomised controlled trial conducted at a specialist NHS outpatient addictions clinics to determine if mental imagery (of future positive [recovery oriented] events) and a visuospatial task (playing Tetris) can help reduce cue-induced alcohol craving. Effects of both interventions will be compared.

DETAILED DESCRIPTION:
Alcohol misuse has a devastating economic impact, with alcohol misuse reportedly costing the UK £20 billion a year. The burden on the health system is also well recognized, with for example, 70% of all admissions to A&E could be linked to alcohol misuse. Meanwhile, the links between alcohol misuse and mental health conditions is well recognized, where the prevalence of patients who have a dual diagnosis of Alcohol Use Disorder (AUD) and another psychiatric condition, is well-established in the literature.

Some cognitive models of substance misuse have also hypothesized about the central role that imagery can have in the initiation and maintenance of addiction. The Elaborated Intrusion (EI) Theory hypothesises that elaborating on alcohol related imagery is integral to the craving experience which ultimately leads to drinking. The EI theory describes craving beginning with an intrusive thought, triggered automatically by external or physiological cues, and associated cognitions. Where these thoughts are pleasurable, the individual will likely elaborate. Elaboration is an effortful cognitive event, where sensory information about the substance is searched for and held in working memory as an image. The theory suggests that during the elaboration process, increasingly rich cues serve to heighten the vividness of consumption imagery, giving acquisition even greater urgency and attentional priority. These images are initially rewarding but as elaboration continues, awareness of somatic deficit and negative affect will occur where the target is not acquired and consumed.

As the elaboration is effortful, the theory proposes that the construction and maintenance of these desire images takes up limited working memory capacity. Therefore, the EI theory suggests that were elaboration is disrupted, through a competing task, craving will reduce.

Tetris has now been tested across craving populations to test the EI theory. Research groups have found that playing Tetris was significantly better than a control condition (watching a loading screen) at reduced self-reported craving for a range of targets. Tetris, therefore appears to be an easily accessible tool to operationalise as a means to interfere with visuo-spatial elaboration during craving for patients.

The researchers who developed the EI theory, hypothesise that familiar, habitual sensory imagery around a desired substance will hold vividness and emotive power that is easily maintained where competing imagery is weak and less meaningful or vivid to the individual. In the researcher's view, this is what explains relapse to alcohol, as competing tasks do not hold sufficient pleasure or reward during craving to engage individuals attention. Therefore, while they may agree with evidence that 'blocking' the elaboration of imagery processes is a useful (and more effective start than other non-imagery based distraction tasks), they hypothesise that a personalised and meaningful image with significant reward feature should outperform a visuo-spatial task, such as Tetris, in blocking the craving processes.

Findings support this, suggesting that personally meaningful aspirational or 'positive' images around abstaining can be effective in reducing urges to use. For example, in piloting 'Functional Imagery Training' (FIT), researchers found that patients who rehearsed multisensory positive goal imagery lost more weight and reduced snacking more than a wait list control group. However, no study has compared this 'positive/motivational image' approach to an alternative visuo-spatial working memory task.

This study has the following aims:

* To determine if visualising a meaningful/positive image reduces craving more than engaging in a non-meaningful visuo-spatial task in alcohol use disorder.
* To determine if the vividness of the positive image generated impacts the efficacy of the imagery intervention.
* To determine the pre-morbid ability of the sample in generating prospective/future imagery.
* To determine if the pre-morbid ability for generating prospective/future images impact the efficacy of the imagery intervention.

Participants will be recruited from specialist NHS outpatient addictions clinics (Wandsworth, Bexley and Lambeth community substance misuse services).

Informed consenting adult participants will be randomised to one of two conditions during a single session research appointment:

1. Tetris then Positive Image
2. Positive Image then Tetris

Participants will undergo a craving induction procedure designed to elicit cue-induced craving. In response to elevated craving, participants will be asked to reduce craving levels using a positive future mental imagery intervention and playing Tetris.

Participants will be fully debriefed and provided time to ask any questions they may have. A craving reduction task will also be offered. Participants will also be asked to identify a named person they can contact if they later feel concerned or distressed. Where required, signposting to support will be offered.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent.
* Engaging in working with a community substance misuse service
* Meets DSM-V criteria for alcohol dependency or abuse, or in early recovery.
* Alcohol is the primary substance of dependence.
* 18 years and older.
* Proficient use of the English language to complete questionnaires and an interview.

Exclusion Criteria:

* Cognitive impairment
* Undergoing detoxification for alcohol
* Presence of a psychotic disorder.
* Recent parasuicidal behaviour (last month).
* High levels of intoxication.
* Severe neurodevelopmental disorder (for example Autism/ADHD) that is deemed to impact on the participants' ability to undertake the interview.
* Organic brain injury, including Korsakoff syndrome.
* Currently participating, or recently participated (last month), in other research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Craving Experience Questionnaire - Strength Version (CEQ-S) Score | Throughout study completion, an average of 1.5 hours
  This is a brief, valid and generic measure of craving/desire based on the Elaborated Intrusion Theory of Desire (Kavanagh et al.,2005) and will be completed; 1) on arrival, 2) following the first cue-induction, 3) following the first condition: the tetris task or positive image, 4) following the second cue-induction, 5) following the second condition: the tetris. The CEQ-S measure comprises of 11 items that capture the intensity, imagery and intrusiveness of craving experiences. In the strength scale, participants are asked to rate their experience on a 0-10 likert scale (0=not at all to 10=extremely). Max score = 110 Min score = 0. Higher scores indicate higher strength of craving.

SECONDARY OUTCOMES:
Clinical Outcomes in Routine Evaluation-Outcome Measure: CORE-10 | Approx. minute 5
  This is a valid, reliable and brief 10-item version of CORE-OM used as a screening tool and outcome measure. Items cover anxiety, depression, trauma, physical problems, functioning and risk to self. CORE-10 was designed to assess global distress, such as symptoms of anxiety, depression, risk to self and associated aspects of life and social functioning. Participants rate their level of agreement to the statement on a five-point likert scale (0-4), ('not at all', 'only occasionally', 'sometimes', 'often' and 'most or all of the time') over the last week. Scores range from 0-40. A score on the CORE-10 of 11-15 is indicative of mild psychological distress, 16-20 is moderate, 21-25 equating moderate to severe and 26 and over indicating severe psychological distress.
Prospective Imagery Task (PIT) | Approx. minute 7
  Participants are asked to form a mental image of negative future scenarios and positive future scenarios. The scenarios are comprised of the subjective probability items used by MacLeod et al. (1996) and include events such as ''You will have a serious disagreement with your friend'' or ''You will do well on your course''. Each image is rated for vividness on a continuous 5-point Likert scale anchored at each point from (1) no image at all; (2) vague and dim; (3) unclear but recognisable; (4) moderately vivid; and (5) very vivid. Holmes and colleagues (2008) have adapted a shortened version on this task using 10 negative future scenarios and 10 positive future scenarios, which shall be adopted here. Scores can range from 0-100. Higher scores indicate greater vividness.
SCID-5-CV (Dependence and remission questionnaire). The structured clinical Interview for Diagnostic and Statistical Manual for Mental Disorders. Clinician Version (DSM-5) | Approx. minute 20
  This is a valid and reliable semi-structured interview guide intended to determine whether an individual meets the criteria for the specified DSM V diagnoses and to measure severity of dependence.
Vividness Rating of Positive Image | Approx. minute 60
  This will be measured via 0-100 scale with participant rating how vivid the imaged image was that they generated. Higher score indicates higher vividness.

CONTACTS AND LOCATIONS:
Overall Officials: John Marsden, Prof, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, Psychology & Neuroscience (IoPPN), King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No